CLINICAL TRIAL: NCT00296959
Title: Anti-Dyskinetic Properties of Topiramate: A Double-Blind, Placebo-Controlled Trial in Patients With Parkinson's Disease and Levodopa-Induced Dyskinesias
Brief Title: Topiramate as a Treatment for Levodopa-Induced Dyskinesia in Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: early termination due to slow recruitment
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MDCTOP2005
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-08

CONDITIONS: Parkinson's Disease
Keywords: Dyskinesia; AMPA receptor antagonists
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Topiramate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: topiramate (drug)

SUMMARY:
A phase II double blind trial to evaluate the effects of the AMPA, glutamte antagonist, topiramate on levodopa-induced dyskinesia in Parkinson's disease

DETAILED DESCRIPTION:
The proposed study is a proof-of-concept, Phase II, randomized, double-blind, placebo-controlled, crossover trial to assess the anti-dyskinetic properties of topiramate in patients with PD and bothersome levodopa-induced dyskinesias.

Patients will be randomized to receive tablets of either placebo or topiramate in a double-blind, crossover design using randomization tables. Following the completion of the first arm of the study and the tapering and washout phases, patients will receive topiramate or placebo in a crossover design for the same treatment duration. The dose of topiramate will be slowly escalated twice each week as tolerated. If a patient cannot tolerate a higher dose, the dose will be reduced to the previously tolerated dose.

Clinical assessments during each arm of the study will include the following:

1. Investigator-rated dyskinesia severity (Levodopa challenge): Anti-parkinsonian medications will be held for 12 hours prior to testing. At the time of the assessment, patients will receive the morning dose of either topiramate or placebo and their usual morning levodopa dose. Patients will be videotaped prior to and following medication administration, and dyskinesia severity will subsequently be rated by a blinded investigator. Levodopa challenges will be conducted before each treatment arm (baseline) and at the completion of each treatment arm.
2. Subject-rated dyskinesia severity: Dyskinesia severity will be rated by the patient using several validated methods (Lang-Fahn Activities of Daily Living Dyskinesia scale, Clinical Global Impression, Unified Parkinson's Disease Rating Scale, and home dyskinesia diaries). Rating scales will be completed at the time of each levodopa challenge and at 2-week intervals. Dyskinesia diaries will be completed for 3 days prior to each levodopa challenge.
3. Assessment of parkinsonism: Parkinsonian disability will be assessed using the UPDRS at the baseline evaluation and at the completion of each treatment arm as well as at each bi-weekly visit.
4. Safety and tolerability assessment: During the course of each titration phase, patients will be assessed in the clinic at 2-week intervals, or sooner if indicated. A general physical examination including blood pressure, pulse, and weight as well as detailed questioning regarding possible adverse events and tolerability will be completed. The Epworth Sleepiness Scale will be completed at each visit. Telephone contact will be made on alternate weeks to assess for the occurrence of adverse events and to discuss titration schedules. Patients will be able to reach a physician at all times via pager in the event of difficulties encountered between scheduled contact times.

In addition, for safety monitoring, laboratory tests including urinalysis, clinical chemistries (sodium, potassium, chloride, bicarbonate, BUN, creatinine), CBC with differential, and liver function tests will be followed. These studies will be evaluated at the beginning and end of each treatment arm and mid-way through each dose escalation phase. A baseline EKG will be obtained, and repeat EKGs will be obtained at the completion of each treatment arm.

Results from this study will aid in the development of a larger Phase III clinical trial.

From the proposed trial, information regarding the anti-dyskinetic efficacy of topiramate will be obtained, and tolerability in the PD patient population will be determined.

ELIGIBILITY:
Inclusion Criteria:

* UK PD Society Brain Bank criteria for the diagnosis of idiopathic PD.
* Patients with stable levodopa-induced dyskinesias present greater than 25% of the day (Unified Parkinson's Disease Rating Scale (UPDRS), item 32, rating > 2) and be moderately to completely disabling (UPDRS item 33, rating > 2).
* All anti-parkinsonian medications must be stable for at least one month prior to study enrollment.

Exclusion Criteria:

* Include prior surgery for PD
* Hoehn and Yahr score of 5 when "off"
* History of nephrolithiasis
* Renal impairment
* Liver disease
* Pregnancy
* Premenopausal females and males not using adequate contraception
* Cognitive impairment (Mini Mental State Exam score less than 24)
* History of glaucoma or seizures
* Use of other antiepileptic drugs
* Amantadine
* Carbonic anhydrase inhibitors
* Digoxin
* Metformin
* Or illicit drugs

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
investigator-rated change in dyskinesia severity from video recordings using Goetz Dyskinesia scale

SECONDARY OUTCOMES:
subject-rated change in dyskinesia severity
subject-rated change in dyskinesia disability
subject-rated parkinsonian disability
investigator-rated parkinsonian disability using UPDRS
tolerability
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Fox, MRCP, PhD, Principal Investigator — UHN, Toronto, Canada
Locations (1):
- Toronto Western Hospital, UHN, Toronto, Ontario, Canada